CLINICAL TRIAL: NCT02957188
Title: Metabolism of Uniformly Labelled 13C Eicosapentaenoic Acid and 13C Arachidonic Acid During Healthy Aging
Brief Title: Metabolism of Omega-3 and Omega-6 During Healthy Aging
Status: Completed | Type: Observational
Sponsor: Université de Sherbrooke (Other)
Collaborators: Healthy Aging Research Network (Network)
Responsible Party: Principal Investigator, Mélanie Plourde, Professor, Université de Sherbrooke
Other Study IDs: 13C EPA and 13C AA metabolism
Record Dates: First submitted 2016-10-24; First posted 2016-11-07 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteers
Keywords: Eicosapentaenoic acid; Arachidonic acid; Metabolism; Healthy aging

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Fasted blood samples were collected before breakfast (baseline) and thereafter at 2 h, 4 h, 6 h, 24 h, 7 d, 14 d, after the tracer intake.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Young: Six young (18-30 yrs old) healthy participants were recruited. The study had three blocks of one month: 13C-EPA follow-up, wash-out and 13C-AA follow-up. Each participant orally consumed a single oral dose of 35 mg of 13C-EPA, and after the wash-out, a 50 mg dose of 13C-AA.
  Interventions: Other: 13C eicosapentaenoic acid and 13C arachidonic acid
- Elderly: Six older (≥ 70 yrs old) healthy participants were recruited. The study had three blocks of one month: 13C-EPA follow-up, wash-out and 13C-AA follow-up. Each participant orally consumed a single oral dose of 35 mg of 13C-EPA, and after the wash-out, a 50 mg dose of 13C-AA.
  Interventions: Other: 13C eicosapentaenoic acid and 13C arachidonic acid

INTERVENTIONS:
Other: 13C eicosapentaenoic acid and 13C arachidonic acid — Each participant orally consumed a single oral dose of 35 mg of 13C-EPA, and after the wash-out, a 50 mg dose of 13C-AA.

SUMMARY:
The purpose of this study is to determine the kinetics of 13C-eicosapentaenoic acid (EPA) and 13C-arachidonic acid (AA) in young and older participants

ELIGIBILITY:
Inclusion Criteria:

* six young (18-30 y old) and six older (≥ 70 y old)
* healthy non medicated participants.

Exclusion Criteria:

* Tobacco,
* malnutrition (assessed from blood albumin, haemoglobin and lipids), -
* participants taking an EPA+DHA supplements or consuming more than 2 fish meals per week,
* severe gastro-intestinal problems,
* medication for diabetes,
* thyroid disease,
* renal failure,
* cancer,
* psychiatric difficulties or depression,
* cardiovascular disease,
* glucose intolerance (>8 mmol/L in fasted samples)
* chronic immune condition or inflammation (CRP > 10 mg/l, white cell count),
* recent major surgery or cardiac event,
* dementia,
* ongoing or past severe drug or alcohol abuse,
* ongoing or past intensive physical training.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Young and elderly healthy participants
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2015-08; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Kinetics of 13C-EPA and 13C-AA | Plasma incorporation of 13C-EPA or 13C-AA was measured from the area under the curve in young and older participants over 28 days post-dose

REFERENCES:
- [Derived] Leveille P, Chouinard-Watkins R, Windust A, Lawrence P, Cunnane SC, Brenna JT, Plourde M. Metabolism of uniformly labeled 13C-eicosapentaenoic acid and 13C-arachidonic acid in young and old men. Am J Clin Nutr. 2017 Aug;106(2):467-474. doi: 10.3945/ajcn.117.154708. Epub 2017 Jun 28. PMID 28659301